CLINICAL TRIAL: NCT06306456
Title: A Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Oral Administration of GH21 Capsules Combined With Osimertinib Mesylate Tablets in Patients With Advanced NSCLC With EGFR Mutations
Brief Title: A Phase Ib/II Clinical Study of GH21 Capsules Combined With Osimertinib Mesylate Tablets in Patients With NSCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Genhouse Bio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GH21C201
Record Dates: First submitted 2024-02-29; First posted 2024-03-12 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-02

CONDITIONS: Non-Small Cell Lung Cancer With EGFR Mutation
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 'GH21+Osimertinib'Group (Experimental): GH21 Capsules Combined with Osimertinib Mesylate Tablets
  Interventions: Drug: GH21; Drug: Tagrisso

INTERVENTIONS:
Drug: GH21 — Oral, 15mg BIW/6mg QD
Drug: Tagrisso — Oral, 80mg QD

SUMMARY:
This study, including phase Ib , phase IIa and phase IIb, aims to evaluate the safety, tolerability, PK profile, efficacy and to determine the RP2D of GH21 capsules combined with Osimertinib mesylate tablets in NSCLC patients with EGFR mutations.

DETAILED DESCRIPTION:
Phase Ib: Classic "3+3" design used for Phase 1b to select the putative RDEs. Four dose groups are preset in phase Ib of this study, which including QD groups and BIW groups. Subjects will be enrolled in parallel cross into the group.

Phase IIa: Two cohorts are preset in this stage, Cohort 1: GH21 RDE1 QD + Osimertinib 80 mg QD, Cohort 2: GH21 RDE2 D1D2-BIW + Osimertinib 80 mg QD, Cohort 1 and Cohort 2 are enrolled in parallel.

Phase IIb: Phase IIb preset 1 cohort. The investigator and sponsor will comprehensively evaluate safety, efficacy, and PK data from Phases Ib and IIa to determine the dose level for Phase IIb.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects or their legal representatives can understand and voluntarily sign the written ICF (before the start of screening and any study procedures);
2. Male or female subjects aged ≥18 years;
3. Advanced NSCLC patients with EGFR mutations confirmed by cytological or histological assessments, and meet the following requirement:

   * Phase Ib： patients with disease progression previously at least treated with third-generation EGFR-TKIs and platinum-containing chemotherapy;
   * Phase IIa and IIb：patients with disease progression previously at least treated with a third-generation EGFR-TKIs (Osimertinib, Furmonertinib Almonertinib etc.).
4. Patients have at least one measurable lesion as defined by RECIST v1.1 (a tumor lesion in the area that has undergone radiotherapy or other loco-regional therapies, is generally not considered as measurable unless there is a disease progression in the lesion);
5. Consent to provide samples for genetic testing;
6. Life expectancy of ≥ 3 months;
7. ECOG PS score of 0-1;
8. The subjects must have adequate organ functions;
9. Male and female of reproductive potential must agree to take reliable contraceptive measures (hormone or barrier methods or abstinence) from signing the ICF until 30 days after the last dose. Pregnancy test results must be negative for female of reproductive potential within 7 days prior to the first dose of the investigational product.

Exclusion Criteria:

1. Subjects who receive any chemotherapy or antitumor biologics within 3 weeks, or antitumor therapies such as radiotherapy and endocrine therapy within 4 weeks prior to the first dose of the investigational product, except for the following:

   * Use of nitrosoureas or mitomycin C within 6 weeks prior to the first dose of the investigational product;
   * Oral administration of fluorouracils, small molecule targeted drugs, and Chinese herbal medicines or Chinese patent medicines with antitumor indications within 5 half-lives or 2 weeks before the first dose of the investigational product (whichever is shorter);
   * Small molecule TKI inhibitors within 5 half-lives or 2 weeks prior to the first dose of the investigational product (whichever is shorter);
   * Local palliative radiotherapy within 2 weeks prior to the first dose of the investigational product;
2. Subjects who have had another investigational new drug or therapy within 4 weeks prior to the first dose of the investigational product;
3. Subjects who have had a major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to the first dose of the investigational product, or require an elective surgery during the study;
4. Subjects who have received strong CYP3A4 inhibitors or inducers and strong P-gp inhibitors or inducers within 2 weeks or within 5 half-lives (whichever is longer) prior to the first dose of the investigational product;
5. Subjects with evidence of the following heart conditions:

   * Acute myocardial infarction, unstable angina pectoris, coronary artery bypass grafting, cerebrovascular accident, or transient ischemic attack within 6 months prior to the first dose of the investigational product;
   * Grade III-IV heart failure diagnosed according to the cardiac function classification of the New York Heart Association at screening;
   * Echocardiography (ECHO) shows the left ventricular ejection fraction (LVEF) ≤ 50% at screening;
   * QT interval corrected by Fridericia method (QTcF) is ≥ 450 ms (male) or ≥ 470 ms (female) at screening;
   * Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg) despite of medication treatment at screening;
6. Subjects with dysphagia, gastrointestinal disorders that affect drug absorption, or other malabsorption conditions, such as intestinal obstruction, Crohn's disease, ulcerative colitis, short bowel syndrome, delayed gastric emptying, or severe gastrointestinal toxicities that have not resolved to Grade 2 or lower prior to the first dose of the investigational product; or subjects are diagnosed with a clinically significant or acute gastrointestinal disease;
7. Subjects with poorly controlled clinical pleural ascites assessed by the investigator;
8. Subjects with active central nervous system metastasis and/or carcinomatous meningitis (e.g., brain metastases accompanied by central nervous system symptoms, including headache, vomiting and dizziness, etc.);
9. Subjects with interstitial pneumonia, or any evidence of clinically active interstitial lung disease within 6 months before the first dose of the investigational product;
10. Subjects with a history of other malignancies (excluding those deemed eligible by the investigator, such as skin squamous cell carcinoma in situ, basal cell carcinoma, and cervical cancer in situ that have been cured and have not relapsed for 5 years; or subjects deemed eligible by the investigator in Phase Ib);
11. Subjects with a history of severe allergies, a history of allergies to Osimertinib, or to multiple drugs;
12. Subjects with hepatitis B virus infection (HBsAg positivity and DNA copies < 100 IU/mL); or hepatitis C virus infection (HCV antibody positivity, and HCV RNA > ULN); or human immunodeficiency virus infection (HIV antibody positivity);
13. Subjects with active infections requiring anti-infective treatment (Grade ≥ 2) or fever > 38°C of unknown etiology within 28 days prior to the first dose of the investigational product;
14. Subjects with any toxicity caused by a previous antitumor therapy that has not resolved to Grade ≤ 1 according to CTCAE 5.0 (except for alopecia, Grade 2 peripheral neuropathy, and/or other Grade ≤ 2 AEs of insignificant safety risks) before the first dose of the investigational product;
15. Female subjects who are pregnant or breastfeeding;
16. Subjects who are not suitable for this study due to any clinical or laboratory abnormalities or other reasons as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities | 2 years
  Incidence of dose limiting toxicities (DLTs) in the dose escalation phase. A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first treatment cycle. (phase Ib)
Number of Participants with Adverse Events | 2 years
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imaging and ophthalmological assessments (phase Ib/ IIa)
Progression-Free Survival (PFS) Based on RECIST 1.1 Criteria | 2 years
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death which occurs first. (phase IIb)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Based on RECIST 1.1 Criteria | 2 years
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR). (phase Ib/IIa/IIb)
Duration of Response (DOR) Based on RECIST 1.1 Criteria | 2 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first. (phase Ib/IIa/IIb)
Disease Control Rate (DCR) Based on RECIST 1.1 Criteria | 2 years
  DCR is defined as the proportion of patients in a clinical trial whose cancer shrinks or remains stable over a certain period.
Overall Survival (OS) | 2 years
  OS is defined as the interval of time between the date of first treatment until death, loss to follow up or termination of the study by the sponsor (phase Ib/IIa/IIb)
Plasma Peak Concentration (Cmax) | 2 years
  Highest observed plasma concentration of GH21 and Osimertinib. (phase Ib/IIa/IIb)
Time to Cmax (Tmax) | 2 years
  Time of highest observed plasma concentration of GH21 and Osimertinib. (phase Ib/IIa/IIb)
Area under the Plasma Concentration-Time Curve (AUC) | 2 years
  Area under the plasma concentration time curve of GH21 and Osimertinib. (phase Ib/IIa/IIb)

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Doctorate, Principal Investigator — （86）021-65115006; Haidan Wang, Doctorate, Study Director — （86）0512-86861608
Locations (6):
- China (6):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang